CLINICAL TRIAL: NCT00065832
Title: Early Interventions for Children With Reading Problems
Brief Title: Reading Problems in Children Living in Urban Areas
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD30995-9; 5R01HD030995 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-04 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2004-10

CONDITIONS: Dyslexia
Keywords: Reading disabilities; Inner-city; Urban
MeSH Terms: conditions — Dyslexia

INTERVENTIONS:
Behavioral: Reading Instruction

SUMMARY:
The first line of defense against reading disabilities is good classroom reading instruction. This study describes how characteristics of students, teachers, and instruction relate to academic achievement in inner-city kindergarten through Grade 4 classrooms.

DETAILED DESCRIPTION:
Recent studies show that the incidence of reading disability can be significantly reduced by improving classroom instruction. Effective reading instruction in the primary grades includes explicit instruction in the alphabetic principle, reading for meaning, and opportunities to practice reading and writing. To learn more about the development of literacy skills in urban settings, students in 17 schools in Houston and Washington, D.C., were followed from kindergarten through Grade 4. Schools were selected based on similar demographics: predominantly African-American student population (95%) and high participation in the federal lunch program (85% to 100%). Each school was provided with grade-appropriate reading programs that focused on phonics and spelling. These programs included direct, integrated, classroom, and individual instruction modules.

Approximately 1400 children and 114 teachers participated each year in this four-year study. The design was cross-sequential so that the majority of teachers in a grade participated for two years. All children participating in regular education were included in the study. Children below the 25th percentile on a standardized reading test were tutored individually by retired teachers, using materials from the classroom reading program. A variety of reading curricula were in place in the classrooms across these two sites. In order to help teachers implement these materials effectively, an ongoing research-based professional development model was employed, with curriculum consultants and coaches working with the teachers in the classroom. Researchers observed in each classroom four to six times during the year using on-the-minute recordings of content. Observers also completed ratings of teaching competencies. Teachers completed surveys of knowledge, experience, attitudes, and instructional strategies. A random selection of eight to ten students were assessed four times during the year for growth in literacy-related skills and once at the end of the year for achievement in reading, spelling, and writing.

ELIGIBILITY:
Inclusion Criteria

* Student in participating school
* Kindergarten through Grade 4

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1400
Dates: Start 1993-07; Study Completion 2002-06

CONTACTS AND LOCATIONS:
Overall Officials: Barbara R. Foorman, Principal Investigator — University of Texas

REFERENCES:
- [Background] Foorman BR, Anthony J, Seals L, Mouzaki A. Language development and emergent literacy in preschool. Semin Pediatr Neurol. 2002 Sep;9(3):173-84. doi: 10.1053/spen.2002.35497. PMID 12350038
- [Background] Fletcher, J.M., Foorman, B.R., Boudousquie, A., Barnes, M., Schatschneider, C., & Francis, D.J. (2002). Assessment of reading and learning disabilities: A research-based, treatment-oriented approach. Journal of School Psychology, 40, 27-63.
- [Background] Rayner K, Foorman BR, Perfetti CA, Pesetsky D, Seidenberg MS. How should reading be taught? Sci Am. 2002 Mar;286(3):84-91. doi: 10.1038/scientificamerican0302-84. No abstract available. PMID 11857904
- [Background] Foorman, B.R., Francis, D.J., Fletcher, J.M., Schatschneider, C., & Mehta, P. (1998). The role of instruction in learning to read: Preventing reading failure in at-risk children. Journal of Educational Psychology, 90, 37-55.
- [Background] Fletcher, J.M., Foorman, B.R., Francis, D.J., & Schatschneider, C. (Winter, 1997). Prevention of reading failure. Insight, 22-23.
- [Background] Foorman, B. R. (Ed.) (2003). Preventing and Remediating Reading Difficulities: Bringing Science to Scale. Timonium, MD: York Press.
- [Background] Foorman BR, Breier JI, Fletcher JM. Interventions aimed at improving reading success: an evidence-based approach. Dev Neuropsychol. 2003;24(2-3):613-39. doi: 10.1080/87565641.2003.9651913. PMID 14561564
- [Background] Foorman, B.R., Chen, D.T., Carlson, C., Moats, L., Francis, D.J., & Fletcher, J. (2003). The necessity of the alphabetic principle to phonemic awareness instruction. Reading and Writing, 16, 289-324.
- [Background] Foorman, B.R., Fletcher, J.M., & Francis, D.J. (2004). Early reading assessment. In W.M. Evers & H.J. Walberg (Eds.), Testing student learning, evaluating teaching effectiveness (pp. 81-125). Stanford, CA: The Hoover Institution.
- [Background] Foorman, B.R., Fletcher, J.M., & Francis, D.J. (1999). Beginning reading is strategic and by design multi-level. Issues in Education: Contributions from Educational Psychology, 5, 65-75.
- [Background] Foorman, B.R., Fletcher, J.M., & Francis, D.J. (1998). Preventing reading failure by ensuring effective reading instruction. In S. Patton & M. Holmes (Eds.), The keys to literacy. Washington, D.C.: Council for Basic Education.
- [Background] Foorman, B.R., Francis, D.J., Beeler, T., Winikates, D., & Fletcher, J.M. (1997). Early interventions for children with reading problems: Study designs and preliminary findings. Learning Disabilities: A Multidisciplinary Journal, 8, 63-71.
- [Background] Foorman, B.R., Francis, D.J., Davidson, K., Harm, M., & Griffin, J. (2004). Variability in text features in six grade 1 basal reading programs. Scientific Studies in Reading, 8(2), 167-197.
- [Background] Foorman, B.R., Francis, D.J., Fletcher, J.M., & Schatschneider, C. (2000). Misrepresentation of research by other researchers. Educational Researcher, 29, 27-37.
- [Background] Foorman, B.R., Francis, D.J., Fletcher, J.M., Schatschneider, C., & Mehta, P. (1998). The role of instruction in learning to read: Preventing reading failure in at-risk children. Journal of Educational Psychology, 90, 37-55. [Reprinted in Wray, D. (Ed.) (2004). Major Themes in Education. London, UK: Routledge.]
- [Background] Foorman, B.R., Francis, D.J., Fletcher, J.M., Winikates, D., & Mehta, P. (1997). Early interventions for children with reading problems. Scientific Studies of Reading, 1(3), 255-276. (Special issue on reading interventions)
- [Background] Foorman, B.R., Francis, D.J, Shaywitz, S.E., Shaywitz, B.A., & Fletcher, J.M. (1997). The case for early reading interventions. In B. Blachman (Ed.), Foundations of reading acquisition and dyslexia: Implications for early intervention (pp. 243-264). Mahwah, NJ: Erlbaum.
- [Background] Foorman, B.R., & Moats, L.C. (2004). Conditions for sustaining research-based practices in early reading instruction. Remedial and Special Education, 25(1), 51-60.
- [Background] Foorman, B.R., & Schatschneider, C. (2003). Measurement of teaching practices during reading/language arts instruction and its relationship to student achievement. In S. Vaughn and K.L. Briggs (Eds.), Reading in the classroom: Systems for observation of teaching and learning (pp. 1-30). Baltimore, MD: Brookes Publishing Co.
- [Background] Foorman, B.R., Schatschneider, C., Fletcher, J.M., Francis, D.J., & Moats, L.C. (2004). The impact of instructional practices in grades 1 and 2 on reading and spelling achievement in high poverty schools. Manuscript under review.
- [Background] Foorman, B., Seals, L., Anthony, J., & Pollard-Durodola, S. (2003). Vocabulary enrichment program for third and fourth grade African American students: Description, implementation, and impact. In B.Foorman (Ed.) Preventing and Remediating Reading Difficulities: Bringing Science to Scale. (pp. 419-441). Timonium, MD: York Press.
- [Background] Foorman, B.R., & Torgesen, J.K. (2001). Critical elements of classroom and small-group instruction promote reading success in all children. Learning Disabilities Research and Practice, 16(4), 202-211.
- [Background] Francis, D.J., Chen, D.T., Foorman, B.R., Wristers, K., Schatschcneider, C., Carlson, C., & Fletcher, J.M. (2004). Sequencing Approaches to Reading Instruction in Grades 1 and 2: An Application of Segmented Growth Models to Longitudinal Crossover Trials. Manuscript submitted.
- [Background] Mehta, P., Foorman, B.R., Branum-Martin, L., & Taylor, W. P. (in press). Literacy as a unidimensional multilevel construct: Validation, sources of influence, and implications in a longitudinal study in grades 1-4. Scientific Studies of Reading.
- [Background] Moats, L.C., & Foorman, B.R. (2003) Measuring teachers' content knowledge of language and reading. Annals of Dyslexia, 53, 23-45.
- [Background] Moats, L.C., & Foorman, B.R. (2004). How quality of writing instruction impacts fourth graders' writing outcomes. Manuscript in preparation.
- [Background] Pollard-Durodola, S., Seals, L.M., & Foorman, B.R. (in press). Vocabulary enrichment project. Baltimore, MD: Brookes Publishing Co.
- [Background] Rayner K, Foorman BR, Perfetti CA, Pesetsky D, Seidenberg MS. How psychological science informs the teaching of reading. Psychol Sci. 2001 Nov;2(2 Suppl):31-74. doi: 10.1111/1529-1006.00004.. PMID 11878018
- [Background] Schatschneider, C., Fletcher, J., Francis, D., Carlson, C., & Foorman, B. (2004). Kindergarten prediction of reading skills: A longitudinal comparative study. Journal of Educational Psychology, 96(2), 265-282.
- [Background] Schatschneider, C., Francis, D.J., Foorman, B.R., & Fletcher, J.M. (1999). The dimensionality of phonological awareness: An application of item response theory. Journal of Educational Psychology, 91, 439-449.
- [Background] Fletcher, J.M., Foorman, B.R., & Shaywitz, S.E., Shaywitz, B.A. (1999). Conceptual and methodological issues in dyslexia research: A lesson for developmental disorders (pp. 271-306). In H. Tager-Flusberg (Ed.), Neurodevelopmental disorders. Cambridge, MA: MIT Press.
- [Background] Fletcher, J., Francis, D., Shaywitz, B., Foorman, B., & Shaywitz, S. (1998). Intelligence testing and the discrepancy model for children with learning disabilities. Learning Disabilities Research and Practice, 13, 186-203.
- [Background] Foorman, B.R. (1995). Research on The Great Debate: Code-oriented versus whole-language approaches to reading instruction. School Psychology Review, 24, 376-392. (Invited article for special issue on research on reading instruction.)
- [Background] Foorman, B.R., Francis, D., Fletcher, J., & Lynn, A. (1996). Relation of phonological and orthographic processing to early reading: Comparing two approaches to regression-based, reading-level-match designs. Journal of Educational Psychology, 88, 639-652.
- [Background] Foorman, B.R., & Schatschneider, C. (1997). Beyond alphabetic reading: Comments on Torgesen's prevention and intervention studies. Journal of Academic Language Therapy, 1(1), 59-65.
- [Background] Schatschneider C, Carlson CD, Francis DJ, Foorman BR, Fletcher JM. Relationship of rapid automatized naming and phonological awareness in early reading development: implications for the double-deficit hypothesis. J Learn Disabil. 2002 May-Jun;35(3):245-56. doi: 10.1177/002221940203500306. PMID 15493321